CLINICAL TRIAL: NCT00745992
Title: Voriconazole Therapeutic Drug Monitoring and CYP2C19 Genetic Polymorphisms in Taiwanese Patients
Brief Title: Voriconazole Blood Level and Liver Metabolizing Enzyme in Taiwanese Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200801019R; NSC 97-2320-B-002 -016 -MY3
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2008-09

CONDITIONS: Invasive Fungal Infections
Keywords: Voriconazole; Antifungal Agents; Invasive fungal infections; Therapeutic drug monitoring; CYP Genetic polymorphism
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fungal infections: 1. Patients with invasive fungal infections; and
  2. Patients who receive PO or IV voriconazole for more than 3 days
  Interventions: Other: Blood drawn (lab data)

INTERVENTIONS:
Other: Blood drawn (lab data) — 1. Check drug blood level 3-5 days after start of drug, treatment failure, occurence of adverse events, or clinically indicated
  2. Check genetic polymorphism of liver enzyme 3-5 days after start of drug
  Other Names: Plasma concentration; Enzyme genetic polymorphism; SNP

SUMMARY:
Voriconazole is an effective antifungal agent and may decrease morbidity and mortality for patients with invasive fungal infections. It is metabolized via liver enzymes. However, these enzymes exhibit different activities in individual patient (genetic polymorphism). Higher proportions of Asians metabolize voriconazole slower than Caucasians and African Americans do. Slower metabolizers may experience dose-associated adverse events more frequently, such as visual disturbances, liver function test abnormalities, and neurological complications. On the other hand, extensive metabolizer or other physiologic conditions may lead to lower blood levels of voriconazole, which may result in treatment failure.

We plan to enroll patient who take voriconazole and examine their liver enzyme activities and blood samples for peak and trough drug levels. We will collect potential factors affecting voriconazole levels, and correlate the levels with the dosing regimen, activity of liver enzyme, occurrence of adverse events, and treatment outcomes. The goal of this study is to determine if monitoring of voriconazole blood levels is necessary in Taiwan.

DETAILED DESCRIPTION:
The incidence of opportunistic, invasive fungal infections has dramatically increased over the past two decades and they cause high morbidity and mortality in a variety of patient populations. Voriconazole, a triazole antifungal agent, has shown in vitro activity against many yeasts and a variety of mold and dermatophyte isolates. Voriconazole can be administered either orally or parenterally. It exhibits good oral bioavailability and wide tissue distribution. Voriconazole is extensively metabolized by the hepatic cytochrome P450 isoenzymes, CYP 2C19, CYP 2C9 and CYP 3A4. The affinity of voriconazole is greatest for isoenzyme CYP 2C19 which exhibits genetic polymorphism with 15-20% of Asian populations being poor/slow metabolizers, whereas the prevalence is much lower (3-5%) amongst Caucasians and African Americans. Studies conducted in Caucasian and Japanese healthy subjects have demonstrated that poor metabolizers have, on average, four times higher voriconazole AUC than homozygous extensive metabolisers, while the AUC of heterozygous extensive metabolizers is two times higher than that of homozygous extensive metabolizers. The most commonly reported adverse events associated with voriconazole use include visual disturbances, liver function test abnormalities, and neurological complications. All of them have been reported to be associated with higher plasma concentrations and / or doses. In term of efficacy, an analysis showed a trend toward worse outcomes in patients with voriconazole plasma concentrations < 0.5 μg/mL although this remains controversial. Since Asians have more CYP 2C19 polymorphism, we expect to see more patients with a wider range of voriconazole plasma concentrations than in previous studies in Caucasian patients. Our study will likely provide stronger evidence in explanation of the relationship between voriconazole plasma concentrations and clinical observations.

We plan to enroll patient who take voriconazole and examine their CYP 2C19 genotypes and plasma samples for peak and trough concentrations. We will collect potential confounding factors affecting voriconazole plasma concentrations, and correlate the concentrations with the dosing regimen, presence or absence of CYP 2C19 polymorphism, occurrence of adverse events, and treatment outcomes. The result of this study will be beneficial in clarify the international debate on controversial issue in the voriconazole plasma concentration monitoring. The ultimate goals of this study is to determine if monitoring of voriconazole plasma concentrations is desired in select patient populations or under certain circumstances in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization patient or ambulatory patients
* Patients with invasive fungal infections
* Patients who take PO/IV voriconazole more than 3 days

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalization patient or ambulatory patients, Patients with invasive fungal infections, Patients who take PO/IV voricoanzole more than 3 days
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Relationship between treatment outcome and voriconazole plasma levels | continuous observation through treatment course

SECONDARY OUTCOMES:
Relationship between voriconazole plasma levels and CYP2C19 polymorphism | 3-5 days after start of IV/PO voriconazole
Relationship between safety and voriconazole plasma levels | Continuous observation through treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Lin, PharmD, MS, Principal Investigator — Graduate Institute of Clinical Pharmacy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Bruggemann RJ, Donnelly JP, Aarnoutse RE, Warris A, Blijlevens NM, Mouton JW, Verweij PE, Burger DM. Therapeutic drug monitoring of voriconazole. Ther Drug Monit. 2008 Aug;30(4):403-11. doi: 10.1097/FTD.0b013e31817b1a95. PMID 18641555